CLINICAL TRIAL: NCT00043511
Title: A Phase I Trial to Evaluate the Safety and Immunogenicity of the HIV-1 pGA2/JS2 Plasmid DNA Vaccine Given Intramuscularly (IM) in HIV-1 Uninfected Adults
Brief Title: Safety of an HIV DNA Vaccine Given to HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 045; 10593 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2002-08-09; First posted 2002-08-12 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Injections, Intramuscular; HIV Seronegativity; Plasmids; Vaccines, DNA; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: pGA2/JS2 Plasmid DNA Vaccine

SUMMARY:
The purpose of this study is to see if the experimental HIV vaccine pGA2/JS2 is safe and is well tolerated at two different doses. Another important purpose of this study is to observe how the immune system responds to the vaccine at different dose levels.

Vaccines are given to people to help their bodies fight infection. The vaccine being tested in this study is a DNA vaccine. The pGA2/JS2 plasmid DNA vaccine instructs the body to make some HIV proteins. These HIV proteins may trigger an immune response. Because only a few of the many proteins HIV needs are made through DNA vaccination, there is no risk of getting HIV from the vaccination. This and other similar DNA vaccines have been tested for safety in mice, rabbits, and monkeys. The vaccine has been well tolerated at doses to be used in this study.

DETAILED DESCRIPTION:
DNA vaccination has induced immune responses in animals to a number of viral, bacterial, and parasite derived antigens. Early clinical experiences with HIV DNA vaccines in humans indicate: 1) the tolerability and short-term safety of DNA at doses up to 5000 mcg in humans are excellent; and 2) there is potential for immunogenicity.

The pGA2/JS2 DNA vaccine is part of a planned prime/boost regimen of a DNA vaccine prime followed by a modified vaccinia Ankara (MVA) vaccine boost. In studies in monkeys, a combination of a DNA vaccine and an MVA vaccine protected the monkeys against disease caused by a monkey virus similar to HIV. The current study is an initial investigation of the safety and immunogenicity of the DNA vaccine given alone. The pGA2/JS2 DNA vaccine expresses gag, protease, reverse transcriptase, env, tat, vpu, and rev.

Participants are randomized to 1 of 2 groups. People in Group A receive either 2 injections of a lower dose (300 mcg) of the DNA plasmid vaccine or the placebo control. People in Group B receive either 2 injections of a higher dose (3000 mcg) of the DNA plasmid vaccine or the control. Group B will be enrolled only if the vaccine is found to be safe and well-tolerated during the initial 2-week evaluation of all participants in Group A. Participants receive vaccinations administered at Months 0 and 2. All vaccinations are administered by intramuscular (IM) injection in an outpatient setting. Participants have about 10 clinic visits during this study, including the screening and injection visits. Participants give blood and urine samples at study visits. They are tested for HIV before entering the study and 4 more times during the study. Women who can become pregnant may undergo up to 3 pregnancy tests during the study period.

ELIGIBILITY:
Inclusion Criteria

Participants may be eligible for this study if they:

* Are between the ages of 18 and 40.
* Are at low risk of HIV infection.
* Have access to a participating study site and are available for follow-up for 12 months.
* Complete a questionnaire to evaluate understanding of the study prior to enrollment.
* Are willing to receive HIV test results.
* Are in good general health.
* Do not have hepatitis B.
* Are HCV antibody negative or, if HCV antibody positive, are HCV PCR negative.
* Have had a negative HIV blood test within 8 weeks prior to enrollment.
* Women of childbearing potential must agree to use acceptable methods of contraception.
* Note: All inclusion criteria must be assessed within 56 days prior to study entry.

Exclusion Criteria

Participants may not be eligible for this study if they:

* Have been immunized against smallpox.
* Have received HIV vaccines or placebo in a previous HIV vaccine trial.
* Have used drugs that interfere with the immune system within the past 6 months.
* Have received blood products within 120 days before HIV screening.
* Have received immunoglobulin within 60 days before HIV screening.
* Have received a live vaccine within 30 days prior to initial study vaccine administration.
* Have used investigational research agents within 30 days prior to initial study vaccine administration.
* Have received a killed vaccine or allergy treatment injections within 14 days of study vaccine administration.
* Are currently taking anti-TB therapy.
* Have a history of serious harmful reactions to vaccines.
* Have a history of immune system disease.
* Have a history of unstable asthma.
* Have a history of type I or type II diabetes.
* Have a history of thyroid disease.
* Have a history of tissue swelling with serious episodes.
* Have a history of high blood pressure.
* Have a history of a bleeding disorder that was diagnosed by a doctor.
* Have active syphilis.
* Have a history of cancer, unless it has been surgically removed and in the opinion of the investigator is not likely to recur during the study period.
* Have a history of a seizure disorder.
* Have had their spleen removed.
* Have mental illness that would interfere with compliance with the protocol.
* Have any other conditions that, in the judgement of the investigator, would interfere with the study.
* Are pregnant or breast-feeding.
* Note: All exclusion criteria must be assessed within 56 days prior to study entry.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mulligan, Study Chair — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - UCSF, Gen. Clinical Research Ctr., Mt. Zion Hosp., San Francisco, California
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Background] Robinson HL, Pertmer TM. DNA vaccines for viral infections: basic studies and applications. Adv Virus Res. 2000;55:1-74. doi: 10.1016/s0065-3527(00)55001-5. No abstract available. PMID 11050940
- [Background] Gurunathan S, Klinman DM, Seder RA. DNA vaccines: immunology, application, and optimization*. Annu Rev Immunol. 2000;18:927-74. doi: 10.1146/annurev.immunol.18.1.927. PMID 10837079
- [Background] Amara RR, Villinger F, Altman JD, Lydy SL, O'Neil SP, Staprans SI, Montefiori DC, Xu Y, Herndon JG, Wyatt LS, Candido MA, Kozyr NL, Earl PL, Smith JM, Ma HL, Grimm BD, Hulsey ML, Miller J, McClure HM, McNicholl JM, Moss B, Robinson HL. Control of a mucosal challenge and prevention of AIDS by a multiprotein DNA/MVA vaccine. Science. 2001 Apr 6;292(5514):69-74. doi: 10.1126/science.1058915. PMID 11393868
- [Background] Ramshaw IA, Ramsay AJ. The prime-boost strategy: exciting prospects for improved vaccination. Immunol Today. 2000 Apr;21(4):163-5. doi: 10.1016/s0167-5699(00)01612-1. No abstract available. PMID 10740236